CLINICAL TRIAL: NCT02164162
Title: Interventional Double Blinded Randomized and Controlled Trial on the Efficacy of a Robotic-assisted Gait Training in Addition to a Conventional Physical Therapy in Parkinson's Disease
Brief Title: Efficacy of a Robotic-assisted Gait Training in Addition to a Conventional Physical Therapy in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Habilita, Ospedale di Sarnico (Other)
Responsible Party: Principal Investigator, Giovanni Taveggia, MD, Habilita, Ospedale di Sarnico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAR06
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, Lokomat, gait training, rehabilitation.
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Participants received 12 sessions of robotic assisted body weight-supported treadmill training on the Lokomat. Training occurred approximately 3 days/ week for 4 weeks, and each training session on the Lokomat lasted 30 minutes. All sessions were supervised by a trained research therapist. All participants started with 40% body weight-support and an initial treadmill speed of 1.5 km/h. Body weight-support was used primarily to facilitate an increase in walking speed; therefore, progression of training across subsequent sessions was standardized by preferentially increasing speed and then unloading body weight-support.
  Speed was increased to a range of 2.2 to 2.5 km/h before body weight-support was decreased. There was an active attempt to enhance the level of training at each session.
  Interventions: Device: Lokomat (Hocoma, Zurich, Switzerland)
- Control group (Active Comparator): Participants received 20 sessions of conventional physiotherapy. Training occurred approximately 5 days/week for 4 weeks, and each training session lasted 1 hour .Patients allocated to the Control Group performed a general exercise program and a conventional gait training with a 5-minute rest between them. The general exercise program consisted in cardiovascular warm-up exercises, muscle stretching exercises, active-assisted or active isometric and isotonic exercises for the main muscles of the trunk and limbs, relaxation exercises, coordination and dual task activities and balance exercises. The conventional gait therapy was based on the proprioceptive neuromuscular facilitation concept (lasting 30 minutes), with rhythmic initiation, slow reversal, and agonistic reversal exercises applied to the pelvic region, each 10 minutes long.
  Interventions: Other: Conventional physical treatment

INTERVENTIONS:
Device: Lokomat (Hocoma, Zurich, Switzerland) — Patients allocated to the Experimental group performed a Robotic Assistested Gait Training by means of the Lokomat. The Lokomat is robotic device set up as an exoskeleton on the lower limbs of the patient. The system uses a dynamic body weight-support system to support he participant above a motorized treadmill synchronized with the Lokomat.
  Arms: Experimental group
Other: Conventional physical treatment — Patients allocated to the Control Group performed a general exercise program and a conventional gait training. The general exercise program consisted in cardiovascular warm-up exercises, muscle stretching exercises, active-assisted or active isometric and isotonic exercises for the main muscles of the trunk and limbs, relaxation exercises, coordination and dual task activities and balance exercises. The conventional gait therapy was based on the proprioceptive neuromuscular facilitation (PNF) concept (lasting 30 minutes), with rhythmic initiation, slow reversal, and agonistic reversal exercises applied to the pelvic region, each 10 minutes long. The same trained therapist treated all the patients in this group and standardized the duration of each part of the treatment.
  Other Names: Control group
  Arms: Control group

SUMMARY:
In Parkinson's disease, gait disturbances represent one of the most disabling motor symptoms, frequently associated with an increased risk of falls, loss of independence and a negative impact on quality of life. In recent years, the interest in automated robotic devices for gait training for Parkinson's Disease patients has grown. With their consistent, symmetrical lower-limb trajectories, robotic devices provide many of the proprioceptive inputs that may increase cortical activation and improve motor function while minimizing the intervention of a therapist. So the main aim of this study will be to analyze, through a clinical and an instrumental evaluation, the effectiveness of a Lokomat gait training in subjects affected by Parkinson's disease in comparison to a ground conventional gait training.

DETAILED DESCRIPTION:
In Parkinson's disease, gait disturbances represent one of the most disabling motor symptoms, frequently associated with an increased risk of falls, loss of independence and a negative impact on quality of life. Patients with Parkinson's Disease, display an abnormal gait pattern (reduced gait speed, shortened stride length, and a longer double-limb support phase) and they are typically unable to generate a proper stride length and to maintain a steady gait rhythm. Therefore, improving gait ability is a primary goal of physical therapy in patients with Parkinson's Disease. Conventional Physiotherapy aimed at enabling patients to maintain their maximum level of activity and independence is often prescribed, but treatments for gait give only limited benefits. Promising reports have suggested that external sensory cueing (acoustic, visual, verbal cues), through an attention mechanism, may help to increase the deficient internal cueing in Parkinson's Disease, thus improving gait pattern.Treadmill training, which induces a constant horizontal movement, generates a rhythmic input for locomotion, coordinating the upper and lower limbs, offering a useful retraining modality that complements conventional therapy. In the last decade some researchers focused on the use of partial body weight support systems on the ground or with the combination of treadmill training (Body weight support-treadmill). These systems, which improves the ability to stand in an upright position with a redistribution of forces on the trunk, thus disengaging the girdle and upper limbs, suggests a greater improvement in motor performance and walking ability compared with conventional phisiotherapy. In recent years, the interest in automated robotic devices for gait training for Parkinson's Disease patients has grown. With their consistent, symmetrical lower-limb trajectories, robotic devices provide many of the proprioceptive inputs that may increase cortical activation and improve motor function while minimizing the intervention of a therapist. Moreover, proprioceptive inputs may share mechanisms that are common to external cues, thus stimulating the cerebellar-premotor pathway to improve gait. Besides,the preprogrammed walking pattern corresponds to normal gait kinematics including: gait cycle timing, inter-limb and inter-joint coordination, appropriate limb loading, and afferent signaling. A recent randomized controlled trial that compared a comprehensive rehabilitative program vis-à-vis robot-assisted gait training has shown that the latter displays some advantages. A pilot, non-controlled study explored the effect of robot-assisted gait training on freezing of gait.Still, despite recent interest in automated locomotion training, there is still very little evidence to support the superiority of this technique over traditional gait training. A computerized gait analysis represents an useful aid to study gait disturbances. The analysis sets objectives and defines quantitative data about gait changes occurred in a patient, in relation to the progression of underlying disease or th effectiveness of treatments administered (medication, surgery or physical). So the main aim of this study will be to analyze, through a clinical and an instrumental evaluation, the effectiveness of a Lokomat gait training in subjects affected by Parkinson's disease in comparison to a ground conventional gait training

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease stage 2 to 3 (calculated in the "on phase") on the Hoehn and Yahr scale
* independent walking
* clinical-pharmacological stabilization until three months before the beginning of the study.

Exclusion Criteria:

* deficits of somatic sensation involving the legs
* vestibular disorders or paroxysmal vertigo
* other neurological, orthopedic or cardiovascular co-morbility
* severe posture abnormalities
* severe-moderate cognitive impairment (Minmental state ≤ 21)
* severe dyskinesia or "on-off"phases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Timed 6 meter walking test | 4 weeks
  Timed 6-meter walking test evaluate the gait speed. Individual walks without assistance 10 meters and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale Disease rating scale motor sub-scores) | 4 weeks
  a scale to assess the motor specific examination for Parkinson's Disease
Functional Independence Measure | 4 weeks
  to assess daily activities functional autonomy
Barthel Index | 4 weeks
  to assess the degree of disability
Tinetti Test | 4 weeks
  to assess balance and gait ability and the falls risk
Parkinson's Disease Questionnaire -39 item | 4 weeks
  to assess quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Casa di Cura Habilita, Ciserano, Bergamo, Italy